CLINICAL TRIAL: NCT05942820
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of BWC0977 in Healthy Adult Volunteers
Brief Title: The Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of BWC0977 in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: CMC challenges
Sponsor: Bugworks Research Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C002-2023-001
Record Dates: First submitted 2023-07-05; First posted 2023-07-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Infectious Diseases; Bacterial Infections
Keywords: Safety; Tolerability; Pharmacokinetics; BWC0977
MeSH Terms: conditions — Communicable Diseases; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized in a 3:1 ratio of BWC0977 and Placebo. The following controls will be employed to maintain the double-blind status of the study Infusion solution containing active drug and placebo will be indistinguishable in appearance Randomization list will be provided to the study center pharmacist for dispensing purposes and kept in the pharmacy, accessible to the pharmacist and authorized personnel only PK results for the interim analyses between cohorts will be presented in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWC0977 (Experimental): MAD Cohorts: Subjects will receive multiple doses of 240mg BID 7 days, 750mg BID 10 days,1250mg BID 10 days and 1000mg TID 10 days BWC0977 via IV infusion over 2 hours in the first 4 cohorts. The dose for the A5 cohort will be determined based on safety and tolerability data from the previous cohorts Up to five dose groups will be studied.
  SAD Cohorts: Subjects will receive single doses of BWC0977 via IV infusion over 2 hours. The planned dose to be studied are 1500mg. Upto 2 cohorts will be studied
  Interventions: Drug: BWC0977
- Placebo (Placebo Comparator): Compounded solution minus BWC0977 The placebo used during this study is 5% Dextrose for injection. SAD Cohorts: Subjects will receive single infusions of placebo (Compounded solution minus BWC0977) over two hours. MAD Cohorts: Subjects will receive multiple infusions of placebo over 2 hours for 7 or 10 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BWC0977 — SAD Cohorts: Double-blind dosing will occur. Six participants will receive single doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort. MAD Cohorts: Double blind dosing will occur. Six participants in each cohort will receive multiple doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort. Dosing will commence on the morning of Day 1. Dosing frequency to be confirmed based on safety, tolerability and PK data from SAD cohorts. Daily dosing will continue for a total of 10 consecutive days.
  Arms: BWC0977
Drug: Placebo — SAD Cohorts: Two participants in each cohort will receive a matching placebo. MAD Cohorts: Two participants in each cohort will receive matching placebo.
  Other Names:
  • Compounded solution minus BWC0977
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1 study is designed to assess the safety, tolerabilty and pharmacokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers. This is a randomized double-blind, placebo-controlled, ascending dose, multi-cohort trial. A total of 56 healthy volunteers are expected to be enrolled into 7 Cohorts. The study will be conducted in two phases: A multiple ascending dose (MAD) phase , followed by A single ascending dose (SAD) phase. In SAD, participants in Cohorts 1 - 2 will receive one dose of BWC0977 or placebo. In MAD, participants in Cohorts 6 - 8 will receive multiple doses of BWC0977 or placebo for 10 consecutive days at a dose deemed safe and tolerable as determined in the preceding SAD Cohorts. In both parts sequential cohorts will be exposed to increasing doses of BWC0977.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be eligible for study participation:

1. Healthy male or female 18 to 55 years of age, inclusive, at time of consent.
2. Body mass index (BMI) ≥ 19.0 and ≤ 30.0 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy without clinically significant abnormalities at the screening visit, Day -1 or Day 1, including:

   1. No findings in Physical examination or vital signs (including temperature, HR, respiratory rate, and blood pressure) that the Investigator determines would interfere with interpretation of study results.
   2. Electrocardiograms (ECGs) without clinically significant abnormalities, including a QTcF interval duration ≤450 msec (for males), and ≤470 msec (for females) obtained as an average from the triplicate screening ECGs after at least 5 minutes in a supine quiet-rest position.
   3. Clinically significant abnormalities in the screening clinical laboratory tests, as determined by the Investigator. Repeat testing could be performed at the Investigator's discretion.
4. Willing and able to provide written informed consent.
5. Agrees to be available for all study visits and cooperate fully with the requirements of the study protocol, including the schedule of events.
6. Willing to refrain from strenuous physical activity that could cause muscle aches or injury, including contact sports, at any time from 4 days prior to admission in the clinical research unit (CRU) until completion of the study (follow-up [FU] visit).
7. Willing to refrain from prescription medications from Screening visit until follow-up; and over-the-counter (OTC) medications, vitamin preparations and other food supplements, from Day -1 up to follow-up.
8. Have suitable venous access for drug administration and blood sampling.
9. If female of child-bearing potential, must agree to and comply with:

   1. Using 1 barrier method (e.g., female condom or male partner using a condom) plus 1 other highly effective method of birth control (e.g., oral contraceptive, implant, injectable, indwelling intrauterine device, vasectomized partner), or double-barrier method (use of a condom by the male partner with use of a diaphragm by the female partner), from signing the consent form until 30 days after last study drug administration, or
   2. Sexual abstinence, for the duration of the study (from signing of consent to FU visit) and for 30 days after last study drug administration, plus
   3. Females of child-bearing potential must also agree not to donate ova or oocytes (ie, human eggs) during the study, and for one menstrual cycle after completion of the study.
   4. To be considered of non-childbearing potential, a female must have either a tubal ligation, hysterectomy, bilateral salpingo-oophorectomy (at least 6 weeks prior to screening), or menopause (last menstruation >12 months and FSH in menopausal range); provision of written documentation is not required for female sterilization and oral confirmation is adequate.
   5. Female participants in same sex relationships do not need to utilize contraception.
10. Male volunteers, if sexually active with a female partner, must agree to and comply with using 1 barrier method of birth control (e.g., male condom) plus 1 other highly effective method of birth control in their partner (e.g., oral contraceptive; implant, injectable, indwelling intrauterine device), or double-barrier method (use of a condom by the male partner with use of a diaphragm by the female partner, or sexual abstinence, and must not donate sperm, for the duration of the study (from signing of consent) and for 90 days after last study drug administration.

To be considered surgically sterile, male participants must have had a vasectomy at least 3 months prior to screening with appropriate documentation of the absence of sperm in the ejaculate.

Male participants in same sex relationships do not need to utilize contraception.

Exclusion Criteria:

Volunteers who meet any of the following criteria will be excluded from the study:

1. Women who are pregnant and/or lactating.
2. History or presence of significant cardiovascular (including QT prolongation, clinically significant hypokalemia, or other proarrhythmic conditions), pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine (including glucose intolerance, diabetes mellitus), immunologic (including asthma or seasonal allergies [that require intermittent use of steroids or other medication]), musculoskeletal (including tendinopathy), dermatologic, or neurological disease (including seizure disorders, psychiatric disorders), including any acute illness or surgery within the past 3 months, as determined by the Investigator to be clinically relevant.
3. A serum creatinine value on Day -1 (check-in) that increased by more than 0.2 mg/Dl (or 15.25 μmol/L) from the Screening value. Note: the serum creatinine test may be repeated prior to confirming exclusion.
4. History of photosensitivity to quinolones.
5. History of known or suspected Clostridium difficile infection.
6. Any condition that necessitated hospitalization within the 3 months prior to Day -1 or is likely to require so during the study.
7. Positive test for HbsAg, anti-HCV antibodies, or antibodies to HIV-1, HIV-2 at screening.
8. Exposure to any prescription medications (small molecules, biologics, and vaccines, including influenza and/or COVID-19 vaccines) or, systemically administered OTC drugs, dietary supplements, or herbal remedies, within 14 days or 5 half-lives (if known), whichever is longer, prior to Day 1 (first dose). Participants should not receive any vaccinations (including influenza and/or COVID-19 vaccines) until after study completion. Discussion between the PI and the Sponsor Medical Monitor is encouraged regarding prior use of any medications during the pre-dose period.

   Note: An exception is made for hormonal contraceptives and a limited amount of paracetamol (a maximum of 4 doses per day of 500-mg paracetamol, and no more than 3 g per week) for the treatment of headache or any other pain.
9. Documented hypersensitivity reaction or anaphylaxis to any medication.
10. Smoker (including tobacco, e-cigarettes, or marijuana) or nicotine user within 1 month prior to dosing and have a negative test for cotinine at check in on Day -1 (may be repeated once, at the discretion of the Investigator, in the instance of a positive result).
11. Positive urine drug/alcohol testing at screening or check-in (Day -1), or history of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where one standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years (may be repeated once per timepoint, at the discretion of the Investigator, in the instance of a positive result).
12. Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrollment.
13. Previous participation in this study or previous participation in another study within 5 half-lives (if known) of the agent, or 30 days, whichever is longer, of Day 1.

    Note: prior participation at any time in non-invasive methodology trials in which no drugs were given is acceptable.
14. Consumption of red wine, Seville oranges, grapefruit, or grapefruit juice, pummelos, other citrus fruits, grapefruit hybrids or fruit juices containing such products from 7 days prior to the first dose of study medication.
15. Employee or family member of an employee of the Sponsor, clinical research unit, or clinical research organization at which the study will be conducted.
16. Unable to cooperate fully with the requirements of the study protocol, including the schedule of events, or likely to be non-compliant with any study requirements.
17. Any disease or condition (medical or surgical) that, by the determination of the Investigator, precludes the subject's participation in the study or would place the subject at risk as a result of participation in the study.

Note: Volunteers should refrain from consumption of any foods containing poppy seeds within 48 hours (2 days) prior to screening and prior to Day -1 to avoid false positive drug screen results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Efforts will be made to randomize approximately equal numbers of males and females to either active or placebo in Part 1 and Part 2 (including both genders).
Enrollment: 4 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs and serious adverse events (SAEs) overall and by intensity (Safety and tolerability). | SAD: Up to 7 days; MAD: Up to 15 days
  This outcome combines the measure of the number of participants experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatment

SECONDARY OUTCOMES:
AUC[0-t] of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Area under the plasma concentration curve from time zero to last time of quantifiable concentration (AUC[0-t]) of BWC0977 following single dose administration
AUC[0-inf]) of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  AUC from time zero to infinity (AUC[0-inf]) of BWC0977 following single dose administration
AUC[0-8], AUC[0-12], AUC[0-24]) of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  AUC from time zero to 8, 12, and 24 hours (AUC[0-8], AUC[0-12], AUC[0-24]) of BWC0977 following single dose administration
Cmax of BWC0977 following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Maximum observed plasma concentration (Cmax) of BWC0977 following single dose administration
Cmax of BWC0977 following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start]
  Maximum observed plasma concentration (Cmax) of BWC0977 following repeat dose administration
Terminal half-life (T1/2) | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Terminal half-life (T1/2) of BWC0977 following single dose administration
Systemic clearance (CL) following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Systemic clearance (CL) of BWC0977 following single dose administration
Systemic clearance (CL) following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start]
  Systemic clearance (CL) of BWC0977 following repeat dose administration
Volume of distribution at steady state (Vdss) following single dose administration | Day 1 pre-dose, 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours post infusion start
  Volume of distribution at steady state (Vdss) of BWC0977 following single dose
Pre-dose (trough) concentration (Cτ) at the end of the dosing interval | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start]
  Pre-dose (trough) concentration (Cτ) at the end of the dosing interval of BWC0977 following repeat dose administration
Observed accumulation ratio following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Observed accumulation ratio (Ro) of BWC0977 following repeat dose administration
Volume of distribution at steady state following repeat dose administration | Day 1 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, and 8 hours post infusion start Days 5, 6, 7, 8, and 9: pre-dose Day 10 pre-dose, 30, 60, 75, and 90 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours post infusion start
  Volume of distribution at steady state (Vdss) of BWC0977 following repeat dose
Amount excreted in urine (Ae) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Amount excreted in urine (Ae) of BWC0977 following repeat dose administration
Amount excreted in urine (Ae) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Amount excreted in urine (Ae) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Fraction of the dose excreted in urine (fe) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Fraction of the dose excreted in urine (fe) of BWC0977 following repeat dose administration
Renal Clearance (CLr) following single dose administration | Day 1 pre-dose, 0-2, 2-4, 4-8, 8-12, and 12-24 hours post infusion start
  Renal Clearance (CLr) of BWC0977 following single dose administration
Renal Clearance (CLr) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 10: 0-8 hours post infusion start
  Renal Clearance (CLr) of BWC0977 following repeat dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Farinola, BSc,BMBS, Principal Investigator — CMAX Clinical Research ,Adelaide, SA, Australia, 5000
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No